CLINICAL TRIAL: NCT01955616
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multiple Dose, Parallel Group Study to Evaluate the Pharmacodynamics, Efficacy and Safety of RM-131 Administered to Patients With Parkinson's Disease and Chronic Constipation Dissatisfied With Current Therapy
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of RM-131 in Patients With Parkinson's Disease & Chronic Constipation
Acronym: MOVE-PD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Motus Therapeutics, Inc. (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM-131-007
Record Dates: First submitted 2013-09-25; First posted 2013-10-07 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease, chronic constipation
MeSH Terms: conditions — Parkinson Disease | interventions — relamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RM-131 (Active Comparator): RM-131 100 µg by subcutaneous injection daily in the morning
  Interventions: Drug: RM-131
- Placebo (Placebo Comparator): by subcutaneous injection daily in the morning
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RM-131
  Other Names: Ghrelin receptor agonist; relamorelin
  Arms: RM-131
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study, called MOVE-PD, is to investigate how individuals with Parkinson's disease (PD) and chronic constipation (CC) respond to RM-131 as compared to placebo. The study will look at how well RM-131 affects the frequency of spontaneous bowel movements over a 14-day period. The study will also evaluate the safety and tolerability of the study drug and evaluate whether the study drug relieves the uncomfortable GI symptoms related to chronic constipation in patients who are unsatisfied with other therapies they have tried for constipation.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent and be willing and able to comply with study procedures.
* Diagnosis of Parkinson's disease
* Diagnosis of chronic constipation (CC), including experiencing constipation for ~12 or more weeks in the preceding 12 months.
* Regular treatment for chronic constipation during the last 6 months, and dissatisfaction with current treatment for CC, after treatment with at least 2 regimens for constipation (see note at end of this section).
* Stable medication history defined as no changes in regimen for at least 2 weeks prior to the baseline period
* Body mass index of 18-40 kg/m2
* Mini-mental status exam (at screening) ≥26
* Female patients must have negative serum or urine pregnancy tests and must not be lactating. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. A vasectomized partner will be allowed as one in conjunction with another single-barrier method.
* Female patients unable to bear children must have this documented in the case report form(i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]). Post-menopausal status will be confirmed by follicle stimulating hormone (FSH) in women less than 60 years of age

Note the following medications are allowed:

* Selective serotonin reuptake inhibitor (SSRI), SNRI, and tricyclic antidepressants are permissible at stable doses. All medications shall be reviewed and dis/approved by the investigator on a case-by-case basis.
* Benzodiazepines are permissible at stable doses
* Stable doses of antacids, NSAIDS, Cox-2 inhibitors, calcium supplements, thyroid replacement, estrogen replacements, low-dose aspirin for cardioprotection, and birth control (but with adequate back up contraception as drug interactions with birth control have not been conducted) are permissible
* Dopamine agonists and amantadine allowed if on a stable dose
* Deep brain stimulation is allowed.

Exclusion Criteria:

* Unable or unwilling to provide informed consent or to comply with study procedures
* Diagnosis of secondary constipation beyond that of Parkinson's disease
* Structural or metabolic diseases that affect the GI system
* Unable to withdraw the following medications 48 hours prior to the baseline period and throughout the study (except as protocol defined rescue medications; see below):

  * Medications that alter GI transit including laxatives, prokinetics, erythromycin, narcotics, and anti-cholinergics (except as protocol defined rescue medications).
  * GABAergic agents
  * Drugs with a low therapeutic index, such as warfarin, digoxin, anti-seizure medications
  * NOTE: Parkinson's disease therapies are allowed. Exceptions for Parkinson's disease medications include:

    * Cogentin (benztopine), Artane (trihexyphenidyl), and apomorphone are excluded
* History of recent major surgery (within 60 days of screening)
* Acute or chronic illness or history of illness, which in the opinion of the Investigator, could pose a threat or harm to the patient or obscure interpretation of laboratory test results or interpretation of study data such as frequent angina, Class III or IV congestive heart failure, moderate impairment of renal or hepatic function, poorly controlled diabetes, etc.
* History of symptomatic orthostatic hypotension or significant history of dizziness
* History of hypersensitivity to mannitol which is an ingredient of both active and placebo study medications
* Any clinically significant abnormalities on screening laboratories or physical examination as determined by the Investigator
* Abnormal 12-lead electrocardiogram (ECG), including evidence of acute myocardial or subendocardial ischemia and clinically significant arrhythmias or conduction abnormalities (including prolonged QTc > 500 msec) or abnormal blood pressure at screening except minor deviations deemed to be of no clinical significance by the Investigator
* Acute GI illness within 48 hours of the baseline period
* History of major GI surgery, except that patients with uncomplicated appendectomy or cholecystectomy are allowed.
* ALT or AST > 1.5 X upper limit of normal (ULN) during screening
* Females who are pregnant or breastfeeding
* History of excessive alcohol use or substance abuse
* Patient or caregiver unable to administer daily SC injections
* Participation in an investigational clinical study within the 30 days prior to dosing in the present study
* Any other reason, which in the opinion of the Investigator, would confound proper interpretation of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Investigate the effects of treatment with RM-131 for 14 days on the frequency of spontaneous bowel movements (SBMs) when administered to patients with Parkinson's Disease (PD) and Chronic Constipation (CC) | Screening through Day 28

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of multiple doses of RM-131 when administered to patients with PD and CC | Screening through Day 28
Effect of RM-131 on stool frequency as measured by complete spontaneous bowel movements, stool consistency, straining, completeness of evacuation, abdominal pain, and global patient reported outcomes of severity of constipation and overall relief. | Screening through Day 28
Assess symptoms of Parkinson's disease using the Unified Parkinson Disease Rating Scale (UPDRS) | Screening through Day 28

OTHER OUTCOMES:
Assess the effect of RM-131 on gastroparesis symptoms | Screening through Day 28
Time to first bowel movement (BM) | Screening through Day 28
Area under the concentration versus time curve of RM-131 will be measured | Screening through Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Pfeiffer, MD, Principal Investigator — Parkinson's Study Group
Locations (13):
- United States (13):
  - University of Southern California, Los Angeles, California
  - Colorado Neurological Institute, Englewood, Colorado
  - University of Florida Ctr for Movement Disorders & Neurorestoration, Gainesville, Florida
  - Emory University, Wesley Woods Health Center, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - University of Iowa Hospitals, Movement Disorders Div, Dept of Neurology, Iowa City, Iowa
  - Michigan State University, East Lansing, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Atlantic Neuroscience, Summit, New Jersey
  - University of Rochester, Rochester, New York
  - University of Toledo Medical Center, Toledo, Ohio
  - Movement Disorders Program & The Parkinson's Center of Oregon, Portland, Oregon
  - University of Pennsylvania, Penn Neurological Institute, Philadelphia, Pennsylvania